CLINICAL TRIAL: NCT00532519
Title: Effectiveness of the Selective Serotonin Reuptake Inhibitor,Citalopram (Cipralex), in Prurigo Nodularis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: horcoop-hmo-ctil
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2007-09

CONDITIONS: Prurigo Nodularis
MeSH Terms: interventions — Citalopram; Dexetimide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: citalopram (cipralex) — 10-20 mg/day, for 12 weeks.

SUMMARY:
Prurigo nodularis (PN) is a common dermatological disorder, manifested as scaly nodules which appear mainly on the extensor surfaces of the limbs. PN may appear secondarily to skin scratching in chronic hepatitis, liver cirrhosis, uremia, hypothyroidism etc. Nevertheless, in many cases no underlying physical disease is present. According to the literature, in fifty percent of the patients there is co-morbidity with depression, anxiety or somatoform disorders.

We hypothesize that a group of these patients may benefit from antidepressant therapy.

ELIGIBILITY:
Inclusion Criteria:

* prurigo nodularis
* age: 18-70 years
* agreed to participate

Exclusion Criteria:

* younger than 18 or older than 70
* pregnant or lactating women
* chronic diseases: cancer, neurological disorders, diseases that are known to be associated with pruritus such as liver cirrhosis, uremia, etc.
* sensitivity to cipralotam
* psychosis, bi-polar disorder, substance addiction, use of antidepressant in the previous year
* use of systemic therapies to prurigo nodularis such as thalidomide, cyclosporine

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: liran horev, md, Principal Investigator — Hadassah Medical Organization; rena cooper-kazaz, md, Principal Investigator — Hadassah Medical Organization
Locations (1):
- : Hadassah Medical Organization,, Jerusalem, Israel